CLINICAL TRIAL: NCT04892693
Title: Talazoparib in Advanced Breast Cancer Patients With Homologous Recombinant Deficiency: A Phase II Clinical and Exploratory Biomarker Study of Talazoparib
Brief Title: Talazoparib in Advanced Breast Cancer Patients With Homologous Recombinant Deficiency
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2009-079-1157
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Breast Cancer
Keywords: homologous recombinant deficiency; biomarker study of talazoparib; talazoparib; germline; BRCA
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Intervention Model Description: Single arm, phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talazoparib (Experimental): ; Talazoparib should be taken orally once daily (ie, continuous daily dosing) at approximately the same time each day (preferably in the morning). Daily dosing of talazoparib can be interrupted for recovery from toxicity for up to 28 days. For interruptions longer than 28 days, treatment at the same or a reduced dose can be considered based on the discretion of the treating physician.
  Interventions: Drug: Talazoparib Oral Capsule

INTERVENTIONS:
Drug: Talazoparib Oral Capsule — - Patients will receive Talazoparib 1 mg orally once daily continuously, with or without food. Laboratory values will be monitored every 4 weeks until progression or unacceptable toxicity. Dose modifications should be made based on the observed toxicity
  Other Names: Single arm; Talazoparib

SUMMARY:
Talazoparib has shown clinical efficacy in breast cancer patients with germline BRCA1 or BRCA2 mutations. Beyond BRCA1 and BRCA2 mutations, it is plausible that talazoparib may have activity in patients with homologous recombination defects (HRD).

DETAILED DESCRIPTION:
BRCA 1/2 plays an essential role in homologous recombination repair and breast cancer patients with BRCA 1/2 germline mutation have homologous recombination defects (HRD). Besides BRCA1 or BRCA2 germline mutation, a proportion of breast cancer is characterized as having HRD through germline mutation, somatic mutation, and epigenetic alteration of other homologous recombination repair (HRR) genes (which includes but are not limited to ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, and RAD54L) (5). It is speculated that tumor with HRD may have clinical benefit from PARP inhibitor. However, the efficacy of talazoparib in advanced breast cancer with HRD is not known. The primary purpose of the present study is to evaluate the efficacy of talazoparib in breast cancer with HRD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥19 years old.
2. Pathologically documented breast cancer that is unresectable or metastatic
3. Tumor with homologous recombination deficiency (HRD) defined by

   * Germline or Somatic BRCA1/2 mutation
   * Homologous recombination repair (HRR) genes mutation
   * HRD detected through RAD51 foci formation functional assay
   * HRR genes: ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, and RAD54L
4. Previously treated with a taxane, unless this treatment was contraindicated (whether in recurrent/metastatic setting or in neoadjuvant/adjuvant setting).
5. Previous treatment with platinum therapy in the advanced or metastatic setting is permitted, provided the patient did not have a progression during the platinum treatment. If the patient was treated with neoadjuvant or adjuvant platinum therapy, at least 6 months of disease-free interval is required after the last dose.
6. Documented radiologic progression (during or after most recent treatment or within 6 months after completing adjuvant therapy).

   - If the patients had relapsed within 6 months after adjuvant therapy, this will be counted as a systemic chemotherapy for advanced or metastatic disease.
7. At least 3 weeks has passed since last chemotherapy treatment
8. At least 2 weeks has passed since last hormone therapy or radiation therapy (including palliative radiation).
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
10. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is not feasible) and is suitable for repeated assessment as per RECIST v.1.1.
11. Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7.0 months after the last dose of study treatment.

    - This study recommend "Copper T intrauterine device" as a highly effective methods of contraception (<1% failure rate)
12. Adequate normal organ and marrow function measured within 28 days prior to administration of study treatment

    * Hemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 75 x 109/L
    * Serum bilirubin ≤ 2.0mg/dL [This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.]
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
    * Adequate renal function: Serum creatinine ≤1.5mg/dL or estimated creatinine clearance >60 mL/min
13. Negative urine pregnancy test within 7 days prior to registration in premenopausal patients.
14. Ability to understand and comply with protocol during study period
15. Patients should sign a written informed consent before study entry

Exclusion Criteria:

1. Prior treatment PARP inhibitor
2. However, if the patient participated in a clinical trial evaluating adjuvant PARP inhibitor, patient is allowed to be included in the present study if the patient recurred 6 months after completing PARP inhibitor. No more than three line of previous systemic chemotherapy, excluding neo-adjuvant and adjuvant chemotherapy. (No limitation on hormone therapy. Hormone therapy is not counted as previous line)
3. If there is a standard treatment available for metastatic breast cancer.
4. History of another primary malignancy except for

   * Malignancy treated with curative intent and with no known active disease ≥3 years
   * contralateral breast cancer
   * Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
5. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled GI disease (e.g., Crohn's disease, ulcerative colitis)
6. History of leptomeningeal carcinomatosis
7. Brain metastases or spinal cord compression.

   - Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
8. active infection or immunocompromised patients including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B , hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).

   - Subjects with simple HBV carrier, a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
9. Patients who have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study agents or their excipients.
10. Female patients who are pregnant or breastfeeding.
11. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | Enrollment to end of treatment up to 2 years
  Defined as a complete response (CR) or partial response (PR) on two consecutive assessments, at least 28 days apart, as determined by investigator assessment using RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | First day of study treatment to the date of disease progression or death due to any cause, whichever came first, assessed up to 2 years
  Defined as the time from the date of first dose administration to the first occurrence of disease progression, as determined by investigator assessment using RECIST v1.1, or death from any cause, whichever occurs first.
Duration of objective response (DOR) | Enrollment to end of treatment up to 2 years
  Defined as the time from first occurrence of a documented objective response to disease progression, as determined by investigator assessment using RECIST v1.1 or death from any cause, whichever occurs first
Clinical benefit rate (CBR) | Enrollment to end of treatment up to 2 years
  Defined as having received CR or PR of any duration or stable disease (SD) ≥ 3 months per RECIST v1.1;
Overall survival (OS) | First day of study treatment to the date of death due to any cause, assessed up to 2 years
  Defined as the time from the date of first dose administration to death from any cause
Safety profile (Treatment-related adverse events as assessed by CTCAE v4.0) | First day of study treatment to end of treatment, assessed up to 2 years
  Number of participants with treatment-related adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No